CLINICAL TRIAL: NCT04830826
Title: A Prospective, National, Multi-center, Non-intervention Real-world Study of Adjuvant Therapy in Early Stage NSCLC With EGFR Mutation-Positive in China
Brief Title: A Real-world Study of Adjuvant Therapy in Early Stage NSCLC With EGFR Mutation-Positive in China
Acronym: ADDRESS
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Clinical Professor, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: D7913C00727
Record Dates: First submitted 2021-03-24; First posted 2021-04-05 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: NSCLC, Stage I; NSCLC, Stage II; NSCLC, Stage III
Keywords: EGFR Mutation; NSCLC; Adjuvant Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Surgeries — Surgeries

SUMMARY:
This study is a prospective, national, multi-center, non-interventional study. The main purpose is to explore the initial adjuvant treatment pattern after radical resection for early-stage NSCLC patients with EGFR Mutation-Positive in the real world. The secondary purpose was to observe the postoperative follow-up treatment pattern and its subgroups (based on different EGFR mutation status and different clinical stages).

DETAILED DESCRIPTION:
About 2,000 eNSCLC patients who received radical resection from about 50 research centers across the country will be included in this study, and will be followed up to 2 years after enrollment according to the actual clinical situation. The analysis method of this study is mainly based on descriptive statistics. The information about the human genetic resources of the subjects to be collected includes: demography, physical examination, WHO fitness status, medical history, smoking history, disease characteristics, surgical information, initial and follow-up adjuvant treatment pattern, laboratory tests, survival status, and adverse events related to gefitinib/osimertinib, serious adverse events/non-severe ADR, measures taken for adverse events, outcome of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed;
2. Newly confirmed EGFR Mutation-Positive NSCLC confirmed by histopathology except for cytology;
3. Receiving or not receiving neoadjuvant treatment before surgery;
4. Patients with stage I-III NSCLC undergo confirmed radical R0 resection;

Exclusion Criteria:

1. Patients who currently or have previously participated in any other anti-tumor clinical studies;
2. Patients with NSCLC who have received any systemic anti-cancer therapy as the main treatment in the past. Cytotoxic therapy, targeted therapy (tyrosine kinase inhibitors or monoclonal antibodies) and immunotherapy included except for the use of neoadjuvant therapy;
3. Patients who have received adjuvant therapy before enrollment.
4. Patients with stage I-III NSCLC whose surgical resection cannot be confirmed.
5. Patients assessed by the investigator as unfit for enrollment, such as neurological disorders or metabolic disorders, physical examination or laboratory examination suspected that the patient has a possible disease, or has contraindications to the use of study drugs, or has treatment-related complications High risk etc.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Continuously enroll all patients with early-stage (stage I-III), histopathologically confirmed, and EGFR mutation-positive NSCLC after R0 resection
Sampling Method: Non-Probability Sample
Enrollment: 1490 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
The distribution of participants with initial adjuvant treatment pattern after radical resection surgery for early-stage NSCLC patients | 2 years
  Descriptive summary statistics ( total number of cases, number of missing cases, frequency, and percentage of each category) were used to describe the distribution of participants with initial adjuvant treatment patterns, including chemical, targeted, combined, or other therapy.
  Set subgroup analysis for different initial adjuvant treatment pattern, including different clinical stages (according to phase I/ Phase II/ stage III) and different EGFR mutation status (19del or 21 L858R);
Time on initial adjuvant treatment | 2 years
  Calculate the time from the start date to the end of initial adjuvant treatment. The total number of cases, number of missing cases, mean, standard deviation, median, 25th and 75th percentiles, minimum and maximum were used for statistical description.
The interval from the date of operation to the start date of initial adjuvant therapy with EGFR-TKI. | 2 years
  Calculate the interval of operation to the adjuvant therapy with EGFR-TKI, which is classified into single-drug therapy and combined therapy. The total number of cases, number of missing cases, mean, standard deviation, median, 25th and 75th percentiles, minimum and maximum were used for statistical description.
Numbers of therapy cycles of initial adjuvant treatment | 2 years
  The patients with chemotherapy were mainly calculated, divided into chemotherapy and targeted combination chemotherapy. The total number of chemotherapy cycles, the number of missing cases, the mean, standard deviation, the median, the 25th and 75th percentiles, the minimum and the maximum were statistically described

SECONDARY OUTCOMES:
The distribution of participants with follow-up treatment pattern after initial adjuvant treatment. | 2 years
  Descriptive summary statistics ( total number of cases, number of missing cases, frequency, and percentage of each category) were used to describe the distribution of participants with follow-up treatment patterns after advanced events evaluated by an investigator, including chemical, targeted, combined, or other therapy.
  Set subgroup analysis for different follow-up treatment pattern including different clinical stages (according to phase I/ Phase II/ stage III) and different EGFR mutation status (19del or 21 L858R);
Time on follow-up treatment | 2 years
  Calculate the time from the start date to the end of follow-up treatment. The results are shown in months, to one decimal place. The total number of cases, number of missing cases, mean, standard deviation, median, 25th and 75th percentiles, minimum and maximum were used for statistical description.
The interval from the date of operation to the start date of the follow-up treatment with EGFR-TKI. | 2 years
  Calculate the interval of operation to the follow-up treatment with EGFR-TKI, which is classified into single-drug therapy and combined therapy. The results are shown in months, to one decimal place. The total number of cases, number of missing cases, mean, standard deviation, median, 25th and 75th percentiles, minimum and maximum were used for statistical description.
Numbers of therapy cycles of follow-up treatment | 2 years
  The patients with chemotherapy of follow-up treatment were mainly calculated, divided into chemotherapy and targeted combination chemotherapy. The total number of chemotherapy cycles, the number of missing cases, the mean, standard deviation, the median, the 25th and 75th percentiles, the minimum and the maximum were statistically described

CONTACTS AND LOCATIONS:
Overall Officials: jianxing He, President, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (51):
- China (51):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital，Capital Medical university, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University People'S Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Cancer Center of Guangzhou Medical university, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital,Sun Yat-sen University, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - The second affiliated hospital of guangxi medical university, Nanning, Guangxi
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Anyang Tumour Hospital, Anyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - Bethune first hospital of jilin university, Changchun, Jilin
  - China-Japan Union Hospital of JiLin University, Changchun, Jilin
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Affiliated Hospital of Chifeng University, Chifeng, Neimenggu
  - The Affliated of Inner Mongolia Medical University, Hohhot, Neimenggu
  - Qilu Hospital of Shandong Yniversity, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - PKUCare Luzhong Hospital, Zibo, Shangdong
  - Shanghai Jiaotong University Medical College Affiliated Ruijin hospital, Shanghai, Shanghai Municipality
  - Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - ZhongShan Hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuang
  - The Affliated of Southwest Medical University, Luzhou, Sichuang
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Sir Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The first affiliated hospital zhejiang university, Hangzhou, Zhejiang
  - The Second Affiliated hospital of Zhejiang University Achool of Medical, Hangzhou, Zhejiang
  - Zhejiang cancer hospital, Hangzhou, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - Shaoxing People's Hospital, Shaoxing, Zhejiang
  - Taizhou Hospita of Zhejiang Province, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided